CLINICAL TRIAL: NCT01102595
Title: A Phase II Open Label Randomised Multicentric Study in Patients With Unresectable Glioblastoma Using Neo-adjuvant Treatment With Two Cycles of Temozolomide Previous Temozolomide Plus Radiation Therapy and Adjuvant Temozolomide vs. Neo-adjuvant Treatment With Two Cycles of Temozolomide Plus Bevacizumab Previous Temozolomide, Bevacizumab and Radiation Therapy and Adjuvant Temozolomide.
Brief Title: Neo-adjuvant Treatment With Temozolomide and Bevacizumab Previous to Temozolomide Plus Radiation Plus Bevacizumab Therapy in Unresectable Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GENOM-009
Record Dates: First submitted 2010-04-01; First posted 2010-04-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Glioblastomas
Keywords: Unresectable/inoperable glioblastomas
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Temozolomide plus Radiation (Experimental): Group 1:
  Neoadjuvant phase: Temozolomide 85 mg/m2/d x 21 days every 28 days for 2 cycles.
  Adjuvant phase: Temozolomide 75 mg/m2/d x 42-49 days with standard radiation therapy (60 Gy).
  Maintenance phase: Temozolomide 150 - 200 mg/m2 d1-d5 q 28d for 6 cycles.
  Interventions: Drug: Temozolomide; Radiation: Standard radiation therapy
- 2: Temozolomide plus Radiation plus Bevacizumab (Experimental): Neoadjuvant phase: Temozolomide 85 mg/m2/d x 21 days every 28 days for 2 cycles + bevacizumab 10 mg/kg every 15 days.
  Adjuvant phase: Temozolomide 75 mg/m2/d x 42-49 days with standard radiation therapy (60 Gy) + bevacizumab 10 mg/kg every 15 days.
  Maintenance phase: Temozolomide 150 - 200 mg/m2 d1-d5 q 28d for 6 cycles.
  Interventions: Drug: Temozolomide; Drug: Bevacizumab; Radiation: Standard radiation therapy

INTERVENTIONS:
Drug: Temozolomide — * Temozolomide 85 mg/m2/d x 21 days every 28 days for 2 cycles.
  * Temozolomide 75 mg/m2/d x 42-49 days
  * Temozolomide 150 - 200 mg/m2 d1-d5 q 28d for 6 cycles.
Drug: Bevacizumab — * 2 cycles + bevacizumab 10 mg/kg every 15 days each two cycles.
  * Bevacizumab 10 mg/kg every 15 days, three dosis.
  Arms: 2: Temozolomide plus Radiation plus Bevacizumab
Radiation: Standard radiation therapy — 42-49 days with standard radiation therapy (60 Gy): 2 Gy per day.

SUMMARY:
In the last 20 years, only temozolomide has obtained indication for the treatment of High-grade glioma (HGG). Temozolomide during and later radiation therapy has doubled one year survival and is the standard treatment for glioblastoma. But 30% of glioblastomas receive only a biopsy as they can't be resected and don't get benefit from this treatment. They and should be treated immediately after the biopsy to prevent neurological deterioration but in spite of this approach they often deteriorate neurologically during radiotherapy. . An effective pre-radiation treatment should improve their prognosis and allow them to complete concomitant radiotherapy and temozolomide treatment. Bevacizumab in recurrent HGG displays 63% of objective responses when combined with irinotecan. But irinotecan is not the most active treatment in this disease.

We propose a phase II, two arms, open label, randomized, multicentric study with 2 cycles of temozolomide before radiation therapy and concomitant temozolomide, in patients with glioblastoma and 'biopsy-only'. Bevacizumab will be added to one arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with glioblastoma, non-resectable, biopsy only. Accepting a craniotomy with resection attempted if an RMN within a period of about 72 hours to confirm that the resection was less than 25% of the tumor and fulfill criterion
2. Measurable disease and contrast uptake ≥ 3 cm in one of its diameters.
3. Stable doses of dexamethasone during the week prior to inclusion.
4. Performance Status ≤ 2.
5. Age ≤ 75 years.
6. MiniMental Status> 25/30.
7. Bartel index > 50%.
8. The surgical incision should be healed prior to randomization. The treatment can be started at 3 weeks of a simple stereotactic biopsy or 4 weeks in case of open biopsy (craniotomy).
9. Maximum baseline MRI performed 4 weeks before starting treatment (acceptance of the MRI done for neuronavegation biopsy as baseline).
10. Adequate bone marrow reserve: neutrophils>2000x109/L, platelets>100x109/L, hemoglobin≥106g/dl.
11. Not received prior treatment with chemotherapy or radiation.
12. Adequate renal function: Creatinine <1.5 ULN of the laboratory performing the analysis.
13. Adequate liver function: Serum bilirubin <1.5/ULN SGOT, SGPT<2.5ULN. Serum alkaline phosphatase<3/ULN.
14. Absence of proteinuria.
15. Effective method of contraception for patients and their partners.
16. Written informed consent
17. Collecting material for a double histological confirmation of diagnosis.

Exclusion Criteria:

1. Prior radiotherapy or chemotherapy for the treatment of glioma.
2. Less than 5 years prior to any invasive neoplasia. Accepted carcinoma in situ of cervix carcinoma or cutaneous vasocelular.
3. Cerebral hemorrhage after biopsy.
4. Pregnancy or lactation.
5. Clinically significant cardiovascular disease: - Myocardial infarction or unstable angina (≤ 6 months before randomization) - Congestive heart failure (CHF) class ≥ II NYHA, New York Heart Association. - Cardiac Arrhythmia uncontrolled despite medication (may include patients with atrial fibrillation often controlled). - Peripheral vascular disease ≥ grade 3 (ie, symptomatic and interfering with everyday activities or specifying repairs or review).
6. Continued use of aspirin> 325 mg / day, currently or recently (within the 10 days prior to randomization).
7. Currently established treatment with therapeutic doses of anticoagulants Coumarin derivatives (courmarina, warfarin) or a week before starting treatment. It allows the administration of heparin for control of Deep Vein Thrombosis (DVT)
8. Patients with PTSD and patients with inflammatory bowel disease, with risk of perforation.
9. HT with values above 150 mmHg systolic pressure of 100 mmHg and diastolic tension is not controllable with standard antihypertensive drugs.
10. Not healed scars, ulcers or recent bone fracture.
11. Bleeding diathesis or coagulopathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-12; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Response Rate | Until the first 9 weeks of treatment
  To determine differences in clinical activity in terms of objective response after 2 cycles of 4 weeks in both treatment arms in inoperable patients with glioblastoma (RANO criteria)

SECONDARY OUTCOMES:
Percentage of patients who finish treatment | 41 weeks
Progression-free survival | the participants will be followed until disease progression by RANO criteria
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 21 weeks
  Assess the toxicity of the combination of the treatment.
  Temozolamide+bevacizumab+radiation Temozolamide+radiation
  After the inclusion of the first 10 patients treated with bevacizumab arm (arm 2)the inclusion will be temporarily interrupted until the last of these patients completed concomitant treatment (radiation, temozolomide, bevacizumab) to check the safety of treatment with analysis of adverse effects and toxicity.
  following the NCIC 3.0 criteria.
Percentage of patients without neurological deterioration before radiation therapy. | 8 weeks
Overall survival | Until death

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Español de Investigacion en Neurooncologia, Madrid, Madrid, Spain